CLINICAL TRIAL: NCT07331181
Title: A Post-Market, Single-arm, Confirmatory Interventional Clinical Investigation to Evaluate the Performance and Safety of INNEA and INNEA AQUA for the Treatment of Cheek and décolletage Wrinkles
Brief Title: Evaluation of Performance and Safety of INNEA and INNEA AQUA for the Treatment of Cheek and décolletage Wrinkles
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Innate srl (Industry)
Collaborators: 1Med (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INNEA-2022
Record Dates: First submitted 2024-07-16; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Wrinkle; Aging
Keywords: wrinkles; aging of the skin; Innea-2022

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Innea (Other): At visit 0 after collecting the required informations tha patients will be treat with INNEA or Innea Aqua.
  Subjects can be treated in one or two of the following areas with one of the two IPs (which will be the same for the three injections planned):
  * Cheek
  * Décolletage Performance will be evaluated by the Investigator using the Lemperle Rating Scale (LRS) for cheek wrinkles at each visit, and the Global Aesthetic Improvement Scale (GAIS) for décolletage wrinkles at each post-treatment assessment. In addition, global aesthetic appearance of the face will be assessed through GAIS by the Investigator. Skin radiance and turgor will be evaluated by Subjects using a 5-Likert scale.
  Interventions: Device: Innea, Innea Aqua

INTERVENTIONS:
Device: Innea, Innea Aqua — INNEA: one syringe contains 2.0 ml of non-pyrogenic gel. The gel is based on the following: sodium hyaluronate 20 mg/ml
  INNEA AQUA: one syringe contains 2.0 ml of non- pyrogenic gel. The gel is based on sodium hyaluronate 25 mg/ml, trehalose

SUMMARY:
A Post-Market, Single-arm, Confirmatory Interventional Clinical Investigation to evaluate the Performance and Safety of INNEA and INNEA AQUA for the treatment of cheek and décolletage wrinkles

DETAILED DESCRIPTION:
Investigational product:

INNEA and INNEA AQUA are CE-marked medical devices indicated for intradermal injections. In particular:

* INNEA is a sterile, biodegradable, isotonic, dermal filler. INNEA consists of high chain (1,0-1,5 x 106 Dalton) hyaluronic acid (HA), obtained from Streptococcus equip bacteria, formulated to a concentration of 20 mg/ml in a physiologic buffer. Each box contains one syringe of INNEA, two 30G 1⁄2" disposable sterile needles reserved for injection of INNEA and a product leaflet.
* INNEA AQUA is a sterile, biodegradable, isotonic, intradermal filler. INNEA AQUA consists of a calibrated mix of medium weight (1200 - 1500 KDalton) HA and a low weight (200 - 400 KDalton), obtained from Streptococcus equi bacteria, formulated to a concentration of 25 mg/ml in a physiologic buffer and trehalose. Each box contains one syringe of INNEA AQUA, two 30G 1⁄2" disposable sterile needles reserved for injection of INNEA AQUA and a product leaflet.

Indications:

in the physiological process of aging of the skin, the effects of which include inspissation of the horny layer (roughness and reduced radiance of the skin) and changes in the elastic fibers of the dermis (wrinkles),

- in the dermal tissue repair process, in cases of scar results following superficial cutaneous trauma (e.g., acne and chickenpox scars).

Study procedure:

This is a post-market confirmatory interventional clinical investigation aimed to enroll adult women requiring correction of cheek and/or décolleté wrinkles. The investigation will be useful to collect INNEA and INNEA AQUA performance/safety evidence.

Each Subject, after signing the Informed Consent Form (ICF), will enter into a screening phase during which the baseline tests will be conducted. If the Investigator is able to organize and perform all tests in the same day, the screening phase and the baseline visit (V0) may coincide, and the patient can be treated immediately after signing the ICF. For each Subject, 5 visits will be planned during which several assessments will be performed as described in the Flowchart.

At V0, the Investigator will collect demographic data (e.g., sex, age, weight), medical history (e.g., history of autoimmune disease, diabetes, etc.), current clinical condition, drug allergy history, and Fitzpatrick phototype (as per clinical practice) of the enrolled Subject.

At V0, according to the instructions for use (IFU), the enrolled patients will be treated with one of the two IPs:

* INNEA, three injections at one week interval.
* INNEA AQUA, three injections at one week interval.

Subjects can be treated in one or two of the following areas with one of the two IPs (which will be the same for the three injections planned):

* Cheek
* Décolletage Performance will be evaluated by the Investigator using the Lemperle Rating Scale (LRS) for cheek wrinkles at each visit, and the Global Aesthetic Improvement Scale (GAIS) for décolletage wrinkles at each post-treatment assessment. In addition, global aesthetic appearance of the face will be assessed through GAIS by the Investigator. Skin radiance and turgor will be evaluated by Subjects using a 5-Likert scale.

After each injection, the Investigator will record Subjects' pain intensity using the Numerical Rating Scale (NRS).

Safety will include assessment of vital signs and evaluation of possible cutaneous reactions at each visit. Adverse events, concomitant medications, and device deficiencies will be monitored during the entire duration of the study.

A 5-point Likert Scale will be used by Subjects to assess patient satisfaction with treatment at EOS visit (V4).

ELIGIBILITY:
Inclusion Criteria:

1. Patient Informed consent form (ICF) signed;
2. Female Subjects between 35 and 65 years old at the time of the signature of ICF;
3. Subjects with at least 2 (shallow wrinkles) on the Lemperle Rating Scale requiring correction of cheek wrinkles and/or subjects requiring correction of décolletage wrinkles;
4. Willingness to follow all study procedures, including attending all site visits, tests and examinations;
5. Agreeing to present at each study visit without make-up;
6. Willingness not to undergo other procedures involving aesthetic correction (e.g., ultrasound-based treatments, biomaterial implant, lifting, botulinum toxin injections, laser or intense pulsed light treatment, bio-stimulating treatment, chemical peeling, dermabrasion, fillers) during the entire study period;
7. Willingness to follow indications to not be exposed to make-up for 12 hours after injection;
8. Willingness to avoid prolonged exposure to sunlight and UV or using saunas or Turkish baths for one week after the injection.

Exclusion Criteria:

* Other - different - clinical conditions of the skin (i.e. rosacea,psoriasis, vitiligo, active eczema, severe scleroderma, severe acne and diagnosticated cancer with/without ongoing antitumor therapy); 2. Infectious or inflammatory processes near the area of intervention; 3. Presence of naevi in the area to be injected; 4. Ongoing use or exposure to benzalkonium chloride solutions; 5. Patients who tend to develop hypertrophic scarring; 6. Patients with a history of autoimmune disease or who are receiving immune therapy; 7. Patients who are known to be hypersensitive to hyaluronic acid; 8. Presence of cutaneous disease on the tested area, as lesions, malformations and recurrent facial/labial herpes; 9. Presence of tendon, bone or muscular implants near the areaof intervention; 10. Ongoing cutaneous allergies; 11. Known hypersensitivity to cheloids; 12. Allergy or contraindications to device components; 13. Allergy or contraindication to one of the components of local anesthetic (patch or cream); 14. Immune system illnesses; 15. Diabetes mellitus or uncontrolled systemic diseases (endocrine, hepatic renal, cardiac, pulmonary, neurological disorder); 16. Problems with coagulation or undergoing anticoagulant therapy; 17. Patients who are using substances that can prolong bleeding(such as aspirin, nonsteroidal anti-inflammatory drugs, and warfarin); 18. Current treatment with anti-inflammatory drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago), drugs able to influence the test results in the investigator opinion; 19. Known drug and/or alcohol abuse; 20. Mental incapacity that precludes adequate understanding or cooperation; 21. Any previous permanent and nonpermanent cutaneous treatment for aesthetic correction (e.g., ultrasound-based treatments, biomaterial implant, lifting, botulinum toxin injections, laser or intense pulsed light treatment, bio-stimulating treatment, chemical peeling, dermabrasion, fillers) within 6 months prior to study inclusion; 22. Active malignant neoplasm of any type, or history of a malignancy (patients with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years before study enrollment are also acceptable); 23. Pregnancy or breastfeeding; 24. COVID-19 vaccination within one month prior to study inclusion; 25. Current participation in a similar study or during the previous 3 months.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Lemperle Rating scale | 1 month after the last injections
  To evaluate the performance of INNEA and INNEA AQUA for the treatment of cheek and décolletage wrinkles after 1 month from the last injection, the lamperle Rating scale will be used:
  - The Lemperle Rating Scale (LRS) will be used to assess cheek wrinkles at V4 (1 month after the 3rd injection) by study product.
GAIS for improvement | One month after the injections
  The Global Aesthetic Improvement Scale (GAIS) scale will be used to assess improvement of décolletage wrinkles at V4 (1 month after the 3rd injection) by study product.

SECONDARY OUTCOMES:
Outcome for performance with Lemperle Rating scale (LRS) | 1 month after the last injections
  1. To evaluate the performance of INNEA and INNEA AQUA for the treatment of cheek wrinkles at each visit and décolletage wrinkles at each post-treatment assessment, the LRS (for cheek wrinkles) at
  each visit. This scale is used because is based on standardized 6-point (0-5) clinical tool used by dermatologists and plastic surgeons to assess the severity of facial wrinkles and folds, aiding in evaluating the effectiveness of injectable fillers and, anti-aging treatments. It measures wrinkles based on depth, ranging from 0 (no wrinkles) to 5 (extremely deep wrinkles/folds). The success is based on the % of improvement in the state of the wrinkles.
Outcome safety: evaluation of adverse events | 1 month after the last injections
  To assess the safety and tolerability of INNEA and INNEA AQUA evaluation of the frequency of adverse events (AEs) and type
Performance with Gais | 1 month after the last injections
  To evaluate the performance of INNEA and INNEA AQUA to improve aesthetic appearance of the face, the GAIS will be used at each post-treatment assessment.
Performance with Likert scale | 1 month after the last injections
  To evaluate the performance of INNEA and INNEA AQUA to improve skin radiance and turgor of cheek and décolletage, a 5- Likert scale will be used at each visit.
Pain intensity evaluation with NRS scale | 1 month after the last injections
  To evaluate pain intensity after injection of INNEA and INNEA AQUA, a Numerical Rating Scale (NRS) will be used at V0, V1, V2.
Patience Satisfaction with Likert | 1 month after the last injections
  To evaluate patient satisfaction with INNEA and INNEA AQUA, a 5- Likert Scale will be used at the end of study (EOS).
Evaluation of performance with Gais, secondary endpoint | 1 month after the injections
  To evaluate the performance of INNEA and INNEA AQUA for the treatment of cheek wrinkles at each visit and décolletage wrinkles at each post-treatment assessment, the Gais at each visit will be used

OTHER OUTCOMES:
Device deficiency | 1 month after the last injections
  Device deficiency/incidents will be monitored at V0, V1, V2.
Evaluation during the duration of the study with diary | 1 month after the last injections
  Concomitant medications and AEs will be monitored during the entire duration of the study through a diary dispensed to patients at V0.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - ASST degli Spedali Civili di Brescia, Brescia, Brescia
  - Humanitas Research Hospital, Rozzano, MI
  - Campus Biomedico, Roma, Roma